CLINICAL TRIAL: NCT02123290
Title: A Proof-of-Concept, Open Label Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of Single Doses of DSM265 in Adult Patients With Acute, Uncomplicated Plasmodium Falciparum or Vivax Malaria Mono-Infection Over a 35-Day-Extended Observation Period
Brief Title: DSM265 Phase IIa Investigation Treating Plasmodium Falciparum or Vivax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Asociacion Civil Selva Amazonica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMV_DSM265_13_02
Record Dates: First submitted 2014-04-15; First posted 2014-04-25 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Plasmodium Falciparum Malaria; Plasmodium Vivax Malaria
Keywords: Plasmodium; falciparum; malaria; vivax; DSM265; pharmacokinetics; adult
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax; Malaria | interventions — DSM265

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plasmodium falciparum (Experimental): Patients with Plasmodium falciparum malaria
  Interventions: Drug: DSM265 400mg; Drug: DSM265 xmg; Drug: DSM265 ymg
- Plasmodium vivax (Experimental): Patients with Plasmodium vivax malaria
  Interventions: Drug: DSM265 400mg; Drug: DSM265 xmg; Drug: DSM265 ymg

INTERVENTIONS:
Drug: DSM265 400mg
Drug: DSM265 xmg — Dose of DSM265 to be determined based on the results of the first cohort
Drug: DSM265 ymg — Dose of DSM265 to be determined based on the results of the second cohort

SUMMARY:
This will be a Proof-of-concept / Phase IIa, open label study to examine the efficacy of DSM265 in uncomplicated Plasmodium vivax and Plasmodium falciparum blood-stage malaria in adult patients. A minimum of two cohorts (20 patients) and a maximum of 6 cohorts (60 patients, 3 dose levels) will be tested. The starting dose of DSM265 for the first P. vivax and P. falciparum cohorts will be 400 mg. This dose is expected to show complete clearance of parasites by microscopy by Day 7 and a decrease in recrudescence rate assessed at Day 14 (success criteria for dose de-escalation and continuation of the study).

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 45kg and 90kg
* Mono-infection of P. falciparum or P. vivax confirmed by:

  1. Fever, or history of fever in the previous 24 hours and,
  2. Microscopically confirmed parasite infection: 1,000 to 35,000 asexual parasite count/µL blood
* Written informed consent
* Able to swallow oral medication
* Able and willing to participate and to comply with the study requirements
* Agree to hospitalisation for at least 72 hours and until malarial parasites are not detected by microscopy on 2 consecutive occasions
* Agree to return to clinic on Day 5 (in addition to the other study days), if by Day 3 malarial parasites have not fallen below level of detection on at least two consecutive occasions. If there are no longer any signs or symptoms of malaria then to be available every 3-4 days for blood sampling for microscopy and Quantitative Polymerase Chain Reaction, and re-hospitalisation for standard treatment in the event of levels being detectable

Exclusion Criteria:

* Signs and symptoms of severe / complicated malaria according to the World Health Organisation Criteria 2010
* Mixed Plasmodium infection
* Severe vomiting, (more than three times in the 24 hours prior to inclusion) or inability to tolerate oral treatment, or severe diarrhoea
* Presence of other serious or chronic clinical condition requiring hospitalisation
* Severe malnutrition
* Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, QTcB or QTcF interval greater than or equal to 450 msec, personal or family history of long QT syndrome, PR interval >200msec; any degree of heart block), respiratory (including active tuberculosis), history of jaundice, hepatic, renal, gastrointestinal, immunological, neurological (including auditory), endocrine including any type of diabetes mellitus (controlled or not), diabetes insipidus, uncontrolled hypo- or hyperthyroidism, endocrine reproductive disorders not requiring concurrent medication, disorders of adrenal function, infectious conditions other than minor skin or soft tissue infections or confirmed lower urinary tract infection, malignancy, psychiatric, history of convulsions or other neurological or psychiatric abnormality; any other disorder or condition that may render the patient unfit for participation or place him/her at increased risk
* Known active Hepatitis A, Hepatitis B or Hepatitis C antibody
* Any antimalarial treatment in the past:

  * a piperaquine-based compound, mefloquine, naphthoquine or sulphadoxine / pyrimethamine in the previous 6 weeks
  * amodiaquine or chloroquine in the previous 4 weeks
  * quinine, halofantrine, lumefantrine-based compounds and any other anti-malarial treatment or antibiotics with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones, and azithromycin) in the past 14 days
  * any herbal products or traditional medicines, in the past 7 days
* Have received antibacterial treatment with known antimalarial activity in the preceding 14 days
* Have received an investigational drug in the 4 weeks prior to screening
* (a) Aspartate Aminotransferase / Alanine Aminotransferase at least twice the upper limit of normal range and total bilirubin is normal (b) Aspartate Aminotransferase / Alanine Aminotransferase more than 1.5 times the upper limit of normal range and total bilirubin is greater than 1 and less than or equal to 1.5 times the upper limit of normal range
* Hemoglobin level less than or equal to 8g/dL
* Total bilirubin greater than 1.5 times the upper limit of normal range
* Serum creatinine levels more than twice the upper limit of normal range
* Female patients must be neither lactating nor pregnant as demonstrated by a negative pregnancy test at screening and pre-dose and must be willing to take measures not to become pregnant during the study period and safety follow-up period (abstinence or oral contraceptives or double barrier contraception, such as male condom, female condom or diaphragm)
* Any prohibited medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adequate Clinical and Parasitological Response rate at Day 14 | Day 14
  Day 14 clinical and parasitological response rate for Plasmodium falciparum and Plasmodium vivax cohorts
Pharmacokinetic parameter for exposure up to 168 hours | Day 0 to 168 hours post-dose
  Area under the plasma concentration vs time curve from time zero up to and including Day 7 (AUC 0-168)
Pharmacokinetic parameter for exposure AUC (0-t) | Day 0 to Day 28
  Area under the plasma concentration vs time curve from time zero to the time of the last measurable concentration post-dose
Area under the plasma concentration vs time curve from time zero to infinity | To Day 28
  Area under the plasma concentration vs time curve from time zero to the infinity. Participants will be followed for 28 days, data will be extrapolated.
Maximum plasma concentration (Cmax) | Day 0 to Day 28
  Pharmacokinetic parameter maximum plasma concentration
Time to reach maximum plasma concentration (tmax) | Day 0 to Day 28
  Pharmacokinetic parameter: Time to reach maximum plasma concentration (tmax)
Terminal half-life (t½) | Day 0 to Day 28
  Pharmacokinetic parameter: Terminal half-life
The plasma concentration at 168hours post-dose (C168h) | Day 7
  Pharmacokinetic parameter C168 hours
The terminal elimination rate constant | Day 0 to 28
  Pharmacokinetic parameter: The terminal elimination rate constant (Lambda z)

SECONDARY OUTCOMES:
Parasite Clearance kinetics | Day 0 to 28
  1. Parasite clearance time
  2. PRR (Parasite reduction rate) and parasitemia half life
  3. Times to microscopic clearance of asexual parasites
     1. Total reduction
     2. 99% reduction
     3. 90% reduction
     4. 50% reduction
  4. Percent reduction in asexual parasites from baseline (microscopically measured) at 24, 48 and 72 hours post-dose
  5. Proportion of aparasitemic patients at 24, 48 and 72 hours post-dose
Endpoints concerning Safety and tolerability of DSM265 in patients | Day 0 to 28
  For P. falciparum and for P. vivax:
  1. Incidence, severity, drug-relatedness, seriousness of adverse events
  2. Laboratory values (biochemistry and haematology)
  3. Vital signs
  4. ECG findings, including heart rate, ECG intervals (PR, QTcB, QTcF), conduction changes or abnormalities
Endpoints concerning gametocytemia | Days 0 to 28
  1. Percent microscopic reduction in gametocytes (stratified by gametocyte status at inclusion) from baseline at
     1. 24 hours after administration of study drug
     2. 72 hours after administration of study drug
  2. Proportion of subjects with gametocytes (stratified by gametocyte status at inclusion)
  3. Area under the curve (AUC) over 14 and 28 days for gametocyte density (stratified by gametocyte status at inclusion)
The effect of DSM265 on signs and symptoms of malaria | Day 0 to Day 28
  1. 28 day Adequate Clinical and Parasitological Response (for P. vivax and P. falciparum)
  2. Kaplan Meier survival analysis for rate of recurrence, recrudescence and new infection over 28 days in comparison to historical controls
Antimalarial pharmacodynamics - minimum parasiticidal concentration, Minimum Inhibitory Concentration, Time and concentration of parasitemia nadir | Day 0 to Day 28
  1. Minimum Parasiticidal Concentration
  2. Minimum Inhibitory Concentration
  3. Time and concentration of parasitemia nadir (if observed)
  4. A model based link between observed pharmacokinetics and observed parasite density over time

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Llanos, Professor, Principal Investigator — Clínica de la Asociación Civil Selva Amazónica
Locations (1):
- Clínica de la Asociación Civil Selva Amazónica, Iquitos, Departamento de Loreto (Amazonía Peruana), Peru

REFERENCES:
- [Derived] Llanos-Cuentas A, Casapia M, Chuquiyauri R, Hinojosa JC, Kerr N, Rosario M, Toovey S, Arch RH, Phillips MA, Rozenberg FD, Bath J, Ng CL, Cowell AN, Winzeler EA, Fidock DA, Baker M, Mohrle JJ, Hooft van Huijsduijnen R, Gobeau N, Araeipour N, Andenmatten N, Ruckle T, Duparc S. Antimalarial activity of single-dose DSM265, a novel plasmodium dihydroorotate dehydrogenase inhibitor, in patients with uncomplicated Plasmodium falciparum or Plasmodium vivax malaria infection: a proof-of-concept, open-label, phase 2a study. Lancet Infect Dis. 2018 Aug;18(8):874-883. doi: 10.1016/S1473-3099(18)30309-8. Epub 2018 Jun 13. PMID 29909069